CLINICAL TRIAL: NCT03872180
Title: A Phase II Evaluation of Bendamustine, Obinutuzumab and Venetoclax in Patients With Untreated Mantle Cell Lymphoma
Brief Title: Bendamustine, Obinutuzumab, and Venetoclax in Patients With Untreated Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Genentech, Inc. (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jonathon Cohen, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00102827; NCI-2018-00995 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4363-18 (Other: Emory University Hospital/Winship Cancer Institute); ML40204 (Other: Genentech, Inc.); P30CA138292 (NIH)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: CCND1 Positive; Mantle Cell Lymphoma; t(11;14) Positive
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; obinutuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax, bendamustine, obinutuzumab (Experimental): Patients receive venetoclax PO on days 1-28 of course 1 and days 1-10 of subsequent courses, bendamustine IV on days 1 and 2, and obinutuzumab IV on days 1, 8, and 15 of course 1 and day 1 of subsequent courses. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Bendamustine; Biological: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Bendamustine — Given IV
  Other Names: SDX-105
Biological: Obinutuzumab — Given IV
  Other Names: GA-101; Gazyva; RO5072759
Drug: Venetoclax — Given PO
  Other Names: ABT-199; GDC-0199; RG7601; Venclexta; RO5537382

SUMMARY:
This phase II trial studies how well bendamustine, obinutuzumab, and venetoclax work in treating patients with mantle cell lymphoma. Drugs used in chemotherapy, such as bendamustine and venetoclax, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as obinutuzumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving bendamustine, obinutuzumab, and venetoclax may work better in treating patients with mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of the combination of bendamustine, obinutuzumab and venetoclax in patients with untreated mantle cell lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate the safety and dose intensity of the combination of bendamustine, obinutuzumab and venetoclax in untreated mantle cell lymphoma.

II. To explore methods of determining molecular remission for patients with untreated mantle cell lymphoma (MCL).

III. To evaluate long-term outcomes including progression-free and overall survival for patients with untreated MCL who receive the combination.

OUTLINE:

Patients receive venetoclax orally (PO) on days 1-28 of course 1 and days 1-10 of subsequent courses, bendamustine intravenously (IV) on days 1 and 2, and obinutuzumab IV on days 1, 8, and 15 of course 1 and day 1 of subsequent courses. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unaccepted toxicity.

After completion of study treatment, patients are followed up at 45-60 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Ability and willingness to comply with the requirements of the study protocol
* Histologic diagnosis of mantle cell lymphoma. This diagnosis must be confirmed at the treating center and patients must have this diagnosis confirmed by at least one of the following criteria:

  * Fluorescent in situ hybridization (FISH) or conventional cytogenetics positive for t(11;14)
  * Cyclin D1 positive by immunohistochemistry
  * Documentation by a hematopathologist at the treating institution that there is pathologic evidence of mantle cell lymphoma if neither criteria above are met
* No previous therapy for diagnosis of lymphoma (note that in patients deemed to be high-risk for tumor lysis syndrome or for rapid clinical deterioration due to symptomatic disease by the investigator, a short course of steroids designed to decrease tumor burden is permitted)
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2
* Hemoglobin ≥ 9 g/dL
* Absolute neutrophil count ≥ 1.5 x 10⁹/L
* Platelet count ≥ 75 x 10⁹/L
* Serum creatinine ≤ 2.0 mg/dL or creatinine clearance ≥ 40 mL/min
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
* Total bilirubin < 1.5 x ULN (or ≤ 3 x ULN for patients with documented Gilbert syndrome)

  * NOTE: Patients with renal or hepatic impairment that is disease-related (ie, hydronephrosis, hepatic involvement) in the opinion of the investigator but who meet all other eligibility criteria may be considered for enrollment in consultation with the investigational new drug (IND) sponsor, Dr. Jonathon Cohen. Documentation of prior adequate renal/hepatic function and clear association with the disease will be required
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 30 days after the last dose of venetoclax or 18 months after the last dose of obinutuzumab, whichever is longer

  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of obinutuzumab. Men must refrain from donating sperm during this same period
  * With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose of obinutuzumab to avoid exposing the embryo
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

* History of other malignancy that could affect compliance with the protocol or interpretation of results

  * Patients with a history of curatively treated basal or squamous cell carcinoma or Stage 1 melanoma of the skin or in situ carcinoma of the cervix are eligible.
  * Individuals in documented remission without treatment for ≥ 2 years prior to enrollment may be included at the discretion of the investigator. Patients with more recently treated low risk prostate cancer, thyroid cancer, or ductal carcinoma in situ (DCIS) who are felt to be at low risk for progression and who are not currently taking any chemotherapy, hormonal therapy or other anti-cancer therapy are eligible. Patients who have been treated and been in remission for < 2 years must be cleared with the study chair prior to initiating study therapy
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results or that could increase risk to the patient, including renal disease that would preclude chemotherapy administration
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment
* Requires the use of warfarin (because of potential drug-drug interactions that may potentially increase the exposure of warfarin)
* Received strong or moderate cytochrome P450 3A (CYP3A) inhibitors or inducers within 7 days of initiating venetoclax. Consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to first dose of venetoclax
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Presence of positive test results for hepatitis B virus (HBV), hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) antibody

  * Patients who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation
  * Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV deoxyribonucleic acid (DNA) is undetectable. These patients must be willing to undergo monthly DNA testing and to remain on hepatitis B prophylaxis during therapy
* Patients with human immunodeficiency virus (HIV) are eligible if they have a cluster of differentiation 4 (CD4) count > 400 and an undetectable viral load. They must be under the care of an infectious disease physician and have no history of an acquired immune deficiency syndrome (AIDS)-defining illness (except lymphoma)
* Receipt of live-virus vaccines within 28 days prior to the initiation of study treatment or need for live-virus vaccines at any time during study treatment
* Pregnant or lactating, or intending to become pregnant during the study

  * Women of childbearing potential must have a negative serum pregnancy test result within 21 days prior to initiation of study drug
* Recent major surgery (within 6 weeks prior to the start of cycle 1, day 1) other than for diagnosis or line placement
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Known allergy to both xanthine oxidase inhibitors (ie, allopurinol) and rasburicase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2026-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon B. Cohen, MD, MS, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Venetoclax, Bendamustine, Obinutuzumab
Started | 23
Completed | 17
Not Completed | 6
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Venetoclax, Bendamustine, Obinutuzumab
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.74 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Response at Completion of Induction Therapy With This Combination
Description: Response will be assessed by positron emission tomography (PET)/computerized tomography (CT) imaging according to the Lugano Classification for response assessment in lymphoma, developed at the 2014 International Conference on Malignant Lymphoma.
Time Frame: Up to 2.5 years from study start
Measure: Count of Participants; unit: Participants
Arm/Group | Venetoclax, Bendamustine, Obinutuzumab
Number analyzed (Participants) | 23
Participants
  Complete Response | 19
  Partial Response | 1
  Stable/Progressive Disease | 3

2. Secondary Outcome: Rate of Minimal Residual Disease (MRD) Negative Complete Response by ClonoSEQ Mantle Cell Lymphoma (MCL) Assay
Description: MRD will be assessed by peripheral blood using the ClonoSEQ assay available from Adaptive Biotechnologies.
Time Frame: Up to 6 years from study start
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Venetoclax, Bendamustine, Obinutuzumab
Number analyzed (Participants) | 23
Percentage of participants | 8.75 [5.58 to 11.92]

3. Secondary Outcome: Overall Response Rate
Description: Will be summarized descriptively.
Time Frame: Up to 6 years from study start
Measure: Count of Participants; unit: Participants
Arm/Group | Venetoclax, Bendamustine, Obinutuzumab
Number analyzed (Participants) | 23
Participants
  Overall Response Rate (ORR) | 20
  Non-Responders | 3

4. Secondary Outcome: Time to Tumor Progression
Description: Will be summarized descriptively.
Time Frame: Up to 6 years from study start
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Venetoclax, Bendamustine, Obinutuzumab
Number analyzed (Participants) | 23
Months | 8.75 [5.58 to 11.92]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Will be described using the Kaplan-Meier methodology. Some patients may undergo consolidative autologous stem cell transplant without evidence of disease progression. This will not be counted against PFS.
Time Frame: Up to 6 years from study start
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Venetoclax, Bendamustine, Obinutuzumab
Number analyzed (Participants) | 23
Months | 7.0 [1.0 to 14.0]

6. Secondary Outcome: Overall Survival
Description: Will be described using the Kaplan-Meier methodology.
Time Frame: Up to 6 years from study start
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Venetoclax, Bendamustine, Obinutuzumab
Number analyzed (Participants) | 23
Percentage of patients
  6-Month Survival | 87.0 [64.8 to 95.6]
  12-Month Survival | 78.3 [55.4 to 90.3]
  24-Month Survival | 58.2 [34.3 to 76.0]
  36-Month Survival | 51.7 [27.9 to 71.1]

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed up to 6 years and serious, and other (not including serious) Adverse Events were assessed up to 2.5 years.
Arm/Group | Venetoclax, Bendamustine, Obinutuzumab
All-Cause Mortality (participants affected / at risk) | 10/23
Serious Adverse Events (participants affected / at risk) | 8/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax, Bendamustine, Obinutuzumab (N=23)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Tumor Lysis Syndrome (Blood and lymphatic system disorders) | 1 (1)
Hemorrhagic Shock (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax, Bendamustine, Obinutuzumab (N=23)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (9)
Alkaline phosphatase increased (Investigations) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 7 (18)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Anxiety (Psychiatric disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chills (General disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 13 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 11 (18)
Dizziness (Nervous system disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Extrapyramidal disorder (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 15 (19)
Fever (General disorders) | 6 (7)
Flu like symptoms (General disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (3)
Headache (Nervous system disorders) | 9 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (6)
Hypertension (Vascular disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (8)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (12)
Infections and infestations - Other, specify (Infections and infestations) | 4 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (7)
Insomnia (Psychiatric disorders) | 5 (5)
Lymphocyte count decreased (Investigations) | 13 (47)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (4)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 19 (24)
Neutrophil count decreased (Investigations) | 6 (7)
Oral pain (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 3 (3)
Papulopustular rash (Infections and infestations) | 3 (4)
Paresthesia (Nervous system disorders) | 2 (2)
Platelet count decreased (Investigations) | 9 (26)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (5)
Social circumstances - Other, specify (Social circumstances) | 3 (4)
Thromboembolic event (Vascular disorders) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 10 (12)
Weight loss (Investigations) | 3 (4)
White blood cell decreased (Investigations) | 5 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/80/NCT03872180/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT03872180/ICF_002.pdf